CLINICAL TRIAL: NCT00066508
Title: A Phase II Study Of PS-341 (VELCADE) In Chemotherapy-Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Bortezomib in Treating Patients With Diffuse Large B-Cell Lymphoma That Is Refractory To Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316254; UCLA-0301090
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have diffuse large B-cell lymphoma that is refractory to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate in patients with chemotherapy-refractory diffuse large B-cell lymphoma treated with bortezomib.
* Determine the safety and tolerability of this drug in these patients.
* Determine the time to disease progression in patients treated with this drug.
* Determine the possible mechanism of resistance to this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 20 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 22-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell lymphoma, meeting criteria for 1 of the following:

  * Relapsed after prior high-dose chemotherapy with stem cell support
  * Relapsed after prior chemotherapy, including at least 1 prior standard non-Hodgkin's chemotherapy regimen, but not a candidate for high-dose chemotherapy with stem cell support
* Measurable disease

  * At least 1 bidimensionally measurable lesion at least 1.5 cm by CT scan
* No primary or secondary CNS lymphoma
* No HIV-related lymphoma
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* Hemoglobin at least 9 g/dL
* Absolute neutrophil count at least 1,000/mm^3

  * No colony-stimulating factors within 4 weeks before obtaining this result
* Platelet count at least 50,000/mm^3

  * No platelet transfusion within 4 weeks before obtaining this result

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* No active hepatitis B or C viral infection

Renal

* Creatinine no greater than 2 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No evidence of acute ischemia or new conduction system abnormalities on EKG
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Sodium greater than 130 mEq/L
* HIV negative
* No ongoing or active infection
* No other concurrent uncontrolled illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic reaction attributable to compounds of similar chemical or biological composition to bortezomib

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Chemotherapy
* At least 4 weeks since prior immunotherapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy
* More than 12 weeks since prior high-dose chemotherapy with hematopoietic stem cell support

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery unless fully recovered

Other

* Recovered from prior therapy
* No other concurrent investigational agents
* No other concurrent investigational or commercial agents or therapies to treat the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-05; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate (combined complete response and partial response)

SECONDARY OUTCOMES:
Safety
Tolerability
Time to disease progression
Possible mechanism of resistance

CONTACTS AND LOCATIONS:
Overall Officials: Sven De Vos, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States